CLINICAL TRIAL: NCT04605497
Title: A Single Center Open-label Randomized Control Pilot Study to Assess the Efficacy of Real-time Continuous Glucose Monitoring in Subjects With Gestational Diabetes to Increase Glucose Time-in-range
Brief Title: Time-in-range Using Continuous Glucose Monitoring Management of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Miyoshi Valent, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00021775
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Gestational Diabetes
Keywords: Female; pregnancy; gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Use of Dexcom G6 real-time CGM to monitor blood glucose levels continually.
  Interventions: Diagnostic Test: Continuous glucose monitoring (CGM)
- Referent Arm (Other): Self-capillary blood glucose monitoring (SCBG) testing 4x/day with blinded CGM every 2 weeks.
  Interventions: Diagnostic Test: Self-Capillary Blood Glucose Monitoring (SCBG)

INTERVENTIONS:
Diagnostic Test: Continuous glucose monitoring (CGM) — Continual use of CGM to monitor blood glucose levels from enrollment through delivery admission & discharge + additional 10 days during postpartum period
  Arms: Intervention Arm
Diagnostic Test: Self-Capillary Blood Glucose Monitoring (SCBG) — Conventional SCBG 4x/day testing (standard care in Oregon; fasting and 1-hour postprandial) with blinded CGM every 2 weeks SCBG 4 times/day until delivery admission 10 days duration with each blinded CGM wear
  Arms: Referent Arm

SUMMARY:
The continual glucose is going to increase time-in-range compared to the standard method in women with gestational diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Singleton pregnancy ≥20 weeks gestation
* Diagnosed with GDM by either 1-step (IADPSG) or 2-Step (Carpenter-Coustan)
* Compatible, validated phone and operating system to support Dexcom G6 CGM App (See Supplementary Table 1) or option to use receiver

Exclusion Criteria:

* Chronic immunosuppression
* Concomitant disease or condition that may compromise patient safety or the ability to complete study tasks including and not limited to: severe mental illness or a diagnosed or suspected eating disorder
* Known allergy to medical grade adhesives
* Pre-gestational diabetes
* Multifetal gestation
* Current alcohol or illicit drug use
* Simultaneous participation in another clinical study with investigational medicinal product(s) that might have an impact on the study objectives.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Average time-in-range over a 24 hour period | From enrollment to10 days after discharge from hospital following delivery

SECONDARY OUTCOMES:
Average time-in-range during waking hours | From enrollment to10 days after discharge from hospital following delivery
Average time-in-range while asleep | From enrollment to10 days after discharge from hospital following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Amy Valent, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States